CLINICAL TRIAL: NCT00898781
Title: Molecular Detection of Circulating Cancer Cells in Breast, Ovarian, Colon and Pancreatic Cancer
Brief Title: Study of Circulating Cancer Cells in Patients With Metastatic Breast, Ovarian, Colon, or Pancreatic Cancer
Status: Terminated | Type: Observational
Why Stopped: Due to poor accrual
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Charles Erlichman, M.D., Mayo Clinic Cancer Center
Other Study IDs: CDR0000582085; P30CA015083 (NIH); MC0744 (Other: Mayo Clinic Cancer Center); 07-006779 (Other: Mayo Clinic IRB)
Record Dates: First submitted 2009-05-09; First posted 2009-05-12 (Estimated); Last update posted 2011-07-19 (Estimated); Status verified 2011-07

CONDITIONS: Breast Cancer; Colorectal Cancer; Ovarian Cancer; Pancreatic Cancer
Keywords: male breast cancer; stage IV breast cancer; stage IV ovarian epithelial cancer; stage IV ovarian germ cell tumor; stage IV pancreatic cancer; stage IV colon cancer; ovarian sarcoma
MeSH Terms: conditions — Breast Neoplasms; Colorectal Neoplasms; Ovarian Neoplasms; Pancreatic Neoplasms; Breast Neoplasms, Male; Carcinoma, Ovarian Epithelial; Colonic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (6):
- Metastatic Breast Cancer
- Metastatic Ovarian Cancer
- Metastatic Pancreatic Cancer
- Metastatic Colon Cancer
- Stage 3 Ovarian Cancer
- Locally Advanced Pancreatic Cancer

SUMMARY:
RATIONALE: Counting the number of circulating cancer cells in samples of blood from patients with metastatic cancer may help doctors find out how much the cancer has spread.

PURPOSE: This research study is looking at the number of circulating cancer cells in patients with metastatic breast cancer, ovarian cancer, colon cancer, or pancreatic cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* To assess frequency of circulating tumor cells (CTCs) in patients with metastatic ovarian, breast, pancreatic, and colon cancers.
* To assess the variability in number of CTCs between patients with the same tumor type.
* To correlate the number of CTCs with extent of tumor burden as measured by tumor markers, imaging, and the number of metastatic sites and proliferation and apoptotic markers.

OUTLINE: Blood samples are collected before treatment and analyzed using molecular detection techniques to detect circulating cancer cells. Samples are assessed by immunofluorescence for markers of proliferation and survival (e.g., EGFR, phosphorylated EGFR, AKT, phosphorylated AKT, cytokeratins, MAPK, Src, and FAK).

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Radiographic or marker evidence of metastatic ovarian, breast, pancreatic, or colon disease
* Hormone receptor status not specified

PATIENT CHARACTERISTICS:

* Menopausal status not specified
* No history of any prior cancer

PRIOR CONCURRENT THERAPY:

* No prior therapy for metastatic disease

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Registration - Inclusion Criteria
  * Radiographic or marker evidence of metastatic ovarian, breast, pancreatic, or colon disease or pre-operative clinically staged 3 ovarian cancer or locally advanced or metastatic pancreatic cancer.
  * Not received prior therapy for metastatic disease.
  Registration - Exclusion Criteria:
  -History of any prior cancer
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2007-11; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Frequency of circulating cancer cells (CTC) | 1 day
Variability in number of CTCs between patients with the same tumor type | 1 day
Correlation of the number of CTCs with extent of tumor burden as measured by tumor markers, imaging, and the number of metastatic sites and proliferation and apoptotic markers | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Charles Erlichman, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States